CLINICAL TRIAL: NCT04280211
Title: Investigation of Vestibular System Influence in Individuals With Chronic Obstructive Pulmonary Disease
Brief Title: Does Vestibular System Effected in Chronic Obstructive Pulmonary Disease Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nimet Sermenli Aydın (Other)
Responsible Party: Sponsor-Investigator, Nimet Sermenli Aydın, Reseach Assisstant, Trakya University
Organization: Trakya University (Other)
Other Study IDs: 061
Record Dates: First submitted 2020-02-06; First posted 2020-02-21 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Vestibular Disorder
Keywords: vestibular dysfunction; COPD; balance
MeSH Terms: conditions — Vestibular Diseases; Pulmonary Disease, Chronic Obstructive | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD Group: Patients who are over 40 years old, diagnosed with COPD
  Interventions: Other: Respiratory Assessment; Other: Vestibular Assessment; Other: Balance Assessment
- Control Group: Healthy adults over 40 years old
  Interventions: Other: Respiratory Assessment; Other: Vestibular Assessment; Other: Balance Assessment

INTERVENTIONS:
Other: Respiratory Assessment — Spirometric measurement
  Other Names: Respiratory Function Test
Other: Vestibular Assessment — Assessment of peripheral vestibular dysfunction, angular vestibule ocular reflex, vestibular dysfunction
  Other Names: Head shake test; Head trust test; Unterberger test
Other: Balance Assessment — Postural stability
  Other Names: Sensory organization test

SUMMARY:
. The main question is whether the vestibular system is affected by COPD. If there is an influence, the second question is what is the relationship between balance and vestibular interaction in COPD patients. A total of 10 COPD patients and 10 healthy adults will include the study. Respiratory functions, vestibular functions and postural stability of participants will be assessed. This research is planned to be carried out as a cross-sectional/descriptive research. It's planned as a pilot study. Comparisons between study and control groups will be made with independent samples t-test for parametric values and Mann Whitney U for non-parametric values.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disorder (COPD) is a common preventable and treatable disease that is characterized by persistent airflow limitation that is usually progressive and associated with an enhanced chronic inflammatory response in the airways and the lung to noxious particles or gases. Hypoxia caused by restrictive airflow is one of the symptoms of COPD. Hypoxia can affect the inner ear and vestibular nuclei. Also, balance impairment can be caused by hypoxia. Previous studies show that balance affected negatively in COPD patients. The aim of this study is to investigate of vestibular system influence in individuals with COPD. A total of 10 COPD patients and 10 healthy adults will include the study. This research is planned to be carried out as a cross-sectional/descriptive research. It's planned as a pilot study. Respiratory functions (respiratory function test), vestibular functions (head shake test, head trust test, unterberger test) and postural stability (sensory organization test) of participants will be assessed.Comparisons between study and control groups will be made with independent samples t-test for parametric values and Mann Whitney U for non-parametric values.

ELIGIBILITY:
For study group

Inclusion Criteria:

* Volunteering to participate in the study
* Diagnosed with COPD

Exclusion Criteria:

* Communication - Coordination problems of patients
* Using medicine which is increasing the risk of fall
* Any neurologic or musculoskeletal disorders which affect mobility and balance
* Loss of hearing

For control group

Inclusion Criteria:

* Volunteering to participate in the study

Exclusion Criteria:

* Communication - Coordination problems of patients
* Using medicine which is increasing the risk of fall
* Any neurologic, musculoskeletal or respiratory disorders which affect mobility and balance
* Loss of hearing

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group will be selected from Respiratory Disease Hospital - (Süreyyapaşa Göğüs Hastalıkları ve Göğüs Cerrahisi Eğitim ve Araştırma Hastanesi) The control group will be invited from the community by announcements.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-02-25 (Estimated); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Vestibular Assessment 1 | After the individuals permission, in first 4 minutes
  Head Shake Test:The head shake test is performed by shaking the head of the patient. The head is rotated at a comfortable range at a frequency of about 2 to 3 Hertz for 10- to 15 seconds. After shaking, the head remains in the center and the eyes of the patient are observed for nystagmus. The head shake test is used to look for signs of dynamic imbalance of vestibular function by evaluating the post-shaking nystagmus.
Balance Assessment | After the individuals permission, in first 20 minutes
  Subjects stands on dual force plates and and their anterior posterior sway recorded in different test conditions.
  1. Eyes open- stable support
  2. Eyes closed- stable support
  3. Eyes open- stable support
  4. Eyes open-Foam surface
  5. Eyes closed-Foam surface
  6. Eyes open-Foam surface
Respiratory Assessment - Spirometry - Forced expiratory volume in 1 s (FEV1) | After the individuals permission, in first 22 minutes
  *We will supply the information of test results from patients' folders.*
  Forced expiratory volume in 1 s (FEV1)
  Spirometry is the term given to the basic lung function -volume, time and flow- tests that measure the air that is expired and inspired. Spirometry is objective and noninvasive.
  Before performing the forced expiration, tidal (normal) breaths can be taken first, then a deep breath taken in while still using the mouthpiece, followed by a further quick, full inspiration.
Respiratory Assessment - Spirometry - Forced vital capacity (FVC) | After the individuals permission, in first 22 minutes
  *We will supply the information of test results from patients' folders.*
  FVC, the maximum amount of air that can be exhaled when blowing out as fast as possible
  Spirometry is the term given to the basic lung function -volume, time and flow- tests that measure the air that is expired and inspired. Spirometry is objective and noninvasive.
  Before performing the forced expiration, tidal (normal) breaths can be taken first, then a deep breath taken in while still using the mouthpiece, followed by a further quick, full inspiration.
Respiratory Assessment - Spirometry - Vital capacity (VC) | After the individuals permission, in first 22 minutes
  *We will supply the information of test results from patients' folders.*
  Vital capacity (VC), the maximum amount of air that can be exhaled when blowing out as fast as possible
  Spirometry is the term given to the basic lung function -volume, time and flow- tests that measure the air that is expired and inspired. Spirometry is objective and noninvasive.
  Before performing the forced expiration, tidal (normal) breaths can be taken first, then a deep breath taken in while still using the mouthpiece, followed by a further quick, full inspiration.
Respiratory Assessment - Spirometry - Peak expiratory flow (PEF) | After the individuals permission, in first 22 minutes
  *We will supply the information of test results from patients' folders.*
  Peak expiratory flow (PEF), the maximal flow that can be exhaled when blowing out at a steady rate
  Spirometry is the term given to the basic lung function -volume, time and flow- tests that measure the air that is expired and inspired. Spirometry is objective and noninvasive.
  Before performing the forced expiration, tidal (normal) breaths can be taken first, then a deep breath taken in while still using the mouthpiece, followed by a further quick, full inspiration.
Respiratory Assessment - Spirometry - Forced expiratory flow (FEF) | After the individuals permission, in first 22 minutes
  *We will supply the information of test results from patients' folders.*
  Forced expiratory flow, also known as mid-expiratory flow; the rates at 25%, 50% and 75% FVC are given
  Spirometry is the term given to the basic lung function -volume, time and flow- tests that measure the air that is expired and inspired. Spirometry is objective and noninvasive.
  Before performing the forced expiration, tidal (normal) breaths can be taken first, then a deep breath taken in while still using the mouthpiece, followed by a further quick, full inspiration.
Respiratory Assessment - Spirometry - •Inspiratory vital capacity (IVC) | After the individuals permission, in first 22 minutes
  *We will supply the information of test results from patients' folders.*
  Inspiratory vital capacity (IVC), the maximum amount of air that can be inhaled after a full expiration
  Spirometry is the term given to the basic lung function -volume, time and flow- tests that measure the air that is expired and inspired. Spirometry is objective and noninvasive.
  Before performing the forced expiration, tidal (normal) breaths can be taken first, then a deep breath taken in while still using the mouthpiece, followed by a further quick, full inspiration.
Vestibular Assessment 2 | After the individuals permission, in first 8 minutes
  Head Trust Test: A brief, high-acceleration head thrust can test vestibular function of all semicircular canals. Depending on the semicircular canal tested, the head is rotated in a different direction. A corrective catch-up saccade is made in case of vestibular hypofunction.
Vestibular Assessment 3 | After the individuals permission, in first 10 minutes
  Unterberger test: Subjects will close their eyes and begin stepping in place for 60 seconds with shoulder at 90 degrees flexion, arms extended forward. The distance will be measured from the start point to end point.

IPD SHARING:
Plan to Share IPD: Undecided